CLINICAL TRIAL: NCT07266116
Title: A Phase Ib/II Clinical Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of TQB2934 for Injection in Subjects With Systemic Light Chain Amyloidosis
Brief Title: Assessment of the Efficacy and Safety of Injectable TQB2934 (Subcutaneous Injection) in Systemic Light Chain Amyloidosis Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Chia Tai Tianqing Pharmaceutical Technology Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2934-Ib/II-01
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-09

CONDITIONS: Systemic Light Chain Amyloidosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2934 injection (Experimental): TQB2934 injection 40 mg and 60 mg During cycles 1-3, medication is administered once a week. From the end of cycles 4-6, medication is administered once every two weeks. For patients who have not achieved complete remission (CR) or have MRD positivity after six cycles of medication, medication is administered once every eight weeks, with a maximum treatment duration of no more than two years
  Interventions: Drug: TQB2934 injection

INTERVENTIONS:
Drug: TQB2934 injection — TQB2934 for injection is a bispecific antibody targeting B-cell maturation antigen (BCMA) and Cluster of Differentiation 3 (CD3). One end binds to the CD3 receptor on the surface of T cells, while the other end binds to BCMA, recruiting T cells to BCMA-positive cells. This can activate T cells, which then release granzyme, perforin, and other enzymes to kill BCMA-positive malignant plasma cells, thereby reducing the level of monoclonal immunoglobulin light chains in the body and delaying further organ damage.

SUMMARY:
This study is a clinical trial aimed at the marketing of TQB2934 for injection. The project plans to enroll 70 subjects, including 13-21 subjects in Phase Ib, to evaluate the safety and preliminary efficacy, pharmacokinetic (PK) characteristics, immunogenicity, and pharmacodynamic (PD) of TQB2934 for injection in subjects with systemic light chain amyloidosis, and to determine the recommended Phase II dose (RP2D). The Phase II plan involves enrolling 49 subjects, aiming to demonstrate that in adult subjects with relapsed/refractory systemic light chain amyloidosis who have previously received treatment with daratumumab and bortezomib, TQB2934 for injection significantly improves the hematological complete response (CR) rate compared to historical controls. The primary endpoint is the optimal hematological CR rate.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily joined this study, signed the informed consent form, and exhibited good compliance;
* Aged 18 to 75 years old, with an Eastern Cooperative Oncology Group (ECOG) score of 0 to 2, and an expected survival of more than 12 weeks;
* Systemic light chain amyloidosis with diagnostic records (i.e., primary light chain amyloidosis);
* Presence of measurable lesions;
* At least one organ involved;
* Have previously received at least one line of systemic treatment, and have experienced disease recurrence or progression after the last line of treatment was ineffective or the duration of response to the last line of treatment was less than 12 months;
* N-terminal pro-B-type natriuretic peptide (NT-proBNP) ≤ 8500 ng/L;
* The corresponding organ function conforms to the protocol requirements;
* Women of childbearing age should agree to use contraception during the study period and for 6 months after its completion; they must have a negative serum pregnancy test within 7 days before enrollment in the study and must be non-lactating subjects; men should agree to use contraception during the study period and for 6 months after its completion.

Exclusion Criteria:

* Diagnosed with other types of amyloidosis, active plasma cell leukemia, multiple myeloma, etc
* Have received allogeneic hematopoietic stem cell transplantation within 1 year prior to the first dose, or have received autologous hematopoietic stem cell transplantation within 12 weeks prior to the first dose;
* Previously received treatment with drugs targeting the same target;
* Within 4 weeks prior to the first dose, the patient has received a cumulative dose of dexamethasone >160 mg or an equivalent dose of other glucocorticoids, or within 3 weeks prior to the first dose, the patient has received targeted therapy, cytotoxic drugs, or any antibody therapy, or within 2 weeks prior to the first dose, the patient has received proteasome inhibitor therapy or radiotherapy, or within 1 week prior to the first dose, the patient has received immunomodulator therapy;
* Those who have received treatment with traditional Chinese patent medicines and simple preparations with clear anti-tumor indications specified in the National Medical Products Administration (NMPA) approved drug instructions within 2 weeks before the first administration;
* Those who have received attenuated live vaccine within 4 weeks before the first dose or plan to receive attenuated live vaccine during the study period;
* Individuals with a history of severe allergies of unknown cause, or known allergies to monoclonal antibody drugs or exogenous human immunoglobulins, or known allergies to the excipients in injectable TQB2934 or pharmaceutical preparations;
* Having had or currently suffering from other malignant tumors within 3 years before the first medication;
* Unresolved toxic reactions above Common Terminology Criteria (CTC) AE Grade 1 caused by any previous treatment;
* Those who have undergone major surgical treatment, significant traumatic injury, or are expected to undergo major surgery during the study treatment period within 4 weeks before the first dose of medication;
* Arterial/venous thromboembolic events occurred within 6 months before the first dose;
* Individuals with a history of abuse of psychotropic drugs who are unable to quit or who have mental disorders;
* Those with unsatisfactory blood pressure control;
* Patients with poorly controlled diabetes;
* Patients who have active or uncontrolled severe bacterial, viral, or systemic fungal infections (≥CTC AE Grade 2 infections) within 4 weeks before the first dose of medication;
* Patients with hepatitis or decompensated liver cirrhosis (Child-Pugh Class B or C);
* Individuals with active tuberculosis, history of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonia, radiation pneumonia requiring treatment, or clinically symptomatic active pneumonia;
* Those who have experienced asthma within 2 years before the first medication or currently suffer from asthma or chronic obstructive pulmonary disease;
* Have had asthma within 2 years before the first medication or currently suffer from asthma;
* Individuals with significant cardiovascular diseases;
* Individuals with a history of immune deficiency, or active autoimmune diseases requiring systemic immunosuppressive therapy, etc
* Subjects deemed unsuitable for enrollment by the researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-12-26 (Estimated); Primary Completion 2029-02 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Numbers of subjects with adverse events (AEs), abnormal laboratory test values, and serious adverse events (SAEs) | Baseline to the end of the study, about 4 years
  The occurrence of all adverse events (AEs), serious adverse events (SAEs), incidence and severity of adverse events (AEs), abnormal laboratory test values, and serious adverse events (SAEs).
The best hematological response evaluated by the Independent Review Committee (IRC) is complete remission (CR) | Baseline to CR，about 1.5 years
  Percentage of subjects who achieved complete hematological remission (CR) after receiving TQB2934 for injection among adult subjects with relapsed/refractory systemic light chain amyloidosis who had previously received treatment with duramycin and bortezomib.

SECONDARY OUTCOMES:
Peak concentration (Cmax) | Pre-dose Cycle 1 day 1/day 8, post dose Cycle 1 day 8/Cycle 3 day 1 2, 6, 24, 48, 72, 120 hours; pre-dose cycle 1 day 15, 22,cycle 2 day 1, cycle 4 day 1, cycle 6 day 1, cycle 12 day 1 and EOT
  Maximum plasma drug concentration.
Immunogenicity incidence rate and its changes over time | pre-dose day 8, cycle 2 day 1, cycle 6 day 1, cycle 12 day 1 and End of Treatment (EOT)
  Immunogenicity incidence rate and its changes over time
Exploring the correlation between soluble BCMA in peripheral blood and the efficacy of TQB2934 | pre-dose cycle 1 day 1, day 8, cycle 2 day 1, cycle 3 day 1, cycle 6 day 1, cycle 12 day 1; post dose cycle 1 day 1/day 8/cycle 3 day 1 6 hours; 56 days after the last administration
  Exploring the correlation between soluble BCMA in peripheral blood and the efficacy of TQB2934
The best hematologic complete remission rate evaluated by researchers | Baseline to CR, about 1.5 years
  The percentage of subjects with complete remission, which is the best hematological response evaluated by researchers.
Best overall hematologic response rate | Baseline to CR/VGPR/PR, about 1.5 years
  Percentage of subjects with best hematologic response of complete remission (CR), very good partial remission (VGPR), and partial remission (PR)
Minimal residual disease (MRD) negative rate | Baseline to MRD negativity, about 1.5 years
  Percentage of subjects achieving MRD negativity.
Duration of hematologic response (DOR) | The first date of PR/ VGPR/ CR to PD/ major organ failure /die, about 1.5 years
  Among subjects with the best hematological response of CR, VGPR, or PR, the time from the date of first achieving PR or higher response to the date of hematological progression, major organ (heart or kidney) failure, or death (from any cause).
Duration of complete hematological remission (DOCR) | The first date of CR to PD/ major organ failure /die, about 1.5 years
  Among subjects with the best hematological response of CR, the time from the date of first achieving CR to the date of hematological progression, major organ (heart or kidney) failure, or death (from any cause).
Cardiac relief rate | Baseline to Cardiac relief, about 1.5 years
  Percentage of subjects who achieve cardiac remission according to the International Society for Transfusion Medicine (ISA) criteria.
Renal remission rate | Baseline to Renal remission, about 1.5 years
  Percentage of subjects achieving renal remission according to International Society of Amyloidosis (ISA) criteria.
Liver response rate | Baseline to liver remission, about 1.5 years
  Percentage of subjects achieving liver remission according to the International Society of Transfusion Medicine (ISA) criteria.
Main organ dysfunction progression-free survival (MOD-PFS) | The first date of initial medication to PD/ major organ failure /die, about 2 years
  The time from the date of initial medication to the date of hematological progression, major organ (heart or kidney) failure, or death (from any cause).
Major Organ Dysfunction-Event-Free Survival (MOD-EFS) | The first date of initial medication to PD/ major organ failure /die, about 2 years
  The time period from the date of initial medication to the date of hematological progression, major organ (heart or kidney) failure, change of treatment regimen due to poor efficacy or intolerance to toxicity, or death (from any cause).
Overall survival (OS) | The first date of initial medication to die, about 2 years
  The time from the date of initial medication to the date of death from any cause

CONTACTS AND LOCATIONS:
Locations (23):
- China (23):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Southwest Hospital, Third Military Medical University (Army Medical University), Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Guangzhou First Municipal People's Hospital, Guangzhou, Guangdong
  - Peking University ShenZhen Hospital, Shenzhen, Guangdong
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Anyang People's Hospital, Anyang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The first hospital of Jilin University, Changchun, Jilin
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xi'an, Shaanxi
  - Qingdao municipal hosptial (group), Qingdao, Shandong
  - Renji Hospital Shanghai Jiaotong University School Of Medicine, Shanghai, Shanghai Municipality
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Chinese Academy of Medical Sciences Hematology Hospital, Tianjin, Tianjin Municipality
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang